CLINICAL TRIAL: NCT02646176
Title: Comparative Effectiveness of Rehabilitation Interventions for Traumatic Brain Injury
Acronym: TBI-CER
Status: Completed | Type: Observational
Sponsor: Jennifer Bogner, PhD, ABPP (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Jennifer Bogner, PhD, ABPP, Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: OhioU
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Inpatient rehabilitation — Inpatient rehabilitation includes activities and interventions provided by occupational, physical, therapeutic recreation and speech therapists, and psychologists.

SUMMARY:
Traumatic brain injury (TBI) is increasingly recognized as a significant public health issue, but the most effective rehabilitation methods have yet to be identified. The Institute of Medicine and the Agency for Healthcare Quality and Research sponsored systematic reviews of evidence for comparative effectiveness of rehabilitation interventions for TBI. Both reviews concluded that substantially more research is needed to identify interventions best suited for different individuals. The practice-based evidence (PBE) approach employed to create the data used in the proposed study was a research method recommended to provide greater clarity, along with use of patient-centered outcomes obtained over a longer period of time than used in previous studies.

The following specific aims will be addressed in the proposed study:

1. Determine the comparative effectiveness of different therapeutic approaches used in inpatient TBI rehabilitation after statistically adjusting for patient need and ability to benefit from various approaches.

   Investigators hypothesize:

   1.1. Patients who receive a greater proportion of therapy time in Advanced Training (versus Standard of Care) will achieve better outcomes than similar patients who receive a lesser proportion of treatment time in Advanced Training.

   1.2. Patients with the greatest initial levels of disability will experience larger effects from Advanced Training therapeutic approaches in comparison to the effects experienced by patients with less disability at admission.

   1.3. Patients who receive a greater proportion of therapy in contextualized treatment (versus decontextualized) will achieve better outcomes than similar patients who receive a lesser proportion of time in contextualized treatment.
2. Determine the comparative effectiveness of difference in the delivery of inpatient rehabilitation therapies, after statistically adjusting for patient need and ability to benefit.

Investigators hypothesize:

2.1 The level of effort that patients are able to apply in treatment moderates the effectiveness of time in treatment.

2.2 Family involvement in treatment is associated with better outcomes.

Data will be drawn from the database established for the TBI Practice-Based Evidence Study (TBI-PBE Study). Data on 2130 persons who received inpatient TBI rehabilitation at any of 10 sites (9 in US, 1 in Canada) were obtained for the study. Detailed longitudinal data were collected prospectively on rehabilitation therapies (with point of care data completed for every clinical encounter), course of recovery, person and injury characteristics and outcomes during and after rehabilitation. Advanced analytic methods (e.g. propensity scores, generalized linear mixed models) will be used to compare the effects of different rehabilitation interventions on outcomes at discharge and during the 9 months following rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Sustained a TBI, defined as damage to brain tissue caused by external force and evidenced by loss of consciousness, post-traumatic amnesia, skull fracture, or objective neurological findings
2. Diagnosed with an International Classification of Diseases (ICD-9-CM) code consistent with the CDC Guidelines for Surveillance of Central Nervous System Injury
3. Receiving inpatient care on a designated brain injury rehabilitation unit of one of the participating rehabilitation facilities
4. Incurred a TBI severe enough to warrant inpatient rehabilitation regardless of other injuries, with TBI being the predominant reason for rehabilitation admission

Exclusion Criteria:

1. None

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study sample was drawn from the population of persons who received inpatient rehabilitation for TBI in North America.
Sampling Method: Probability Sample
Enrollment: 2130 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Participation | 9 months post-discharge from inpatient rehabilitation
  Participation as measured by the Participation Assessment with Recombined Tools-Objective
Participation | 3 months post-discharge from inpatient rehabilitation
  Participation as measured by the Participation Assessment with Recombined Tools-Objective

SECONDARY OUTCOMES:
Functional independence-Cognitive | Upon completion of inpatient rehabilitation (discharge score), an average of 1 month
  FIM-TM Cognitive scales will be used to measure functional independence in the cognitive realm.
Functional independence-Cognitive | 3 months after discharge from inpatient rehabilitation
  FIM-TM Cognitive scales will be used to measure functional independence in the cognitive realm.
Functional independence-Cognitive | 9 months after discharge from inpatient rehabilitation
  FIM-TM Cognitive scales will be used to measure functional independence in the cognitive realm.
Functional independence-Motor | Upon completion of inpatient rehabilitation (discharge score), an average of 1 month
  FIM-TM Motor scales will be used to measure functional independence in the cognitive realm.
Functional independence-Motor | 3 months post-discharge from inpatient rehabilitation
  FIM-TM Motor scales will be used to measure functional independence in the cognitive realm.
Functional independence-Motor | 9 months post-discharge from inpatient rehabilitation
  FIM-TM Motor scales will be used to measure functional independence in the cognitive realm.
Depressive symptoms | 3 months post-discharge from inpatient rehabilitation
  The Patient Health Questionnaire-9 will be used to measure depressive symptoms.
Depressive symptoms | 9 months post-discharge from inpatient rehabilitation
  The Patient Health Questionnaire-9 will be used to measure depressive symptoms.
Life satisfaction | 3 months post-discharge from inpatient rehabilitation
  The Satisfaction with Life Scale will be used to measure life satisfaction
Life satisfaction | 9 months post-discharge from inpatient rehabilitation
  The Satisfaction with Life Scale will be used to measure life satisfaction
Participation | 3 months post-discharge
  Participation will be measured using the Participation Assessment with Recombined Tools-Objective

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Bogner, PhD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: Yes
A complete de-identified dataset will be made available to the public within 9 months of completion of the analysis.